CLINICAL TRIAL: NCT05901545
Title: Evaluating 111In Panitumumab for Nodal Staging in Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Eben Rosenthal, Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC-EDHAN23201P; NCI-2023-03821 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Panitumumab; Indium; Surgical Procedures, Operative; acetyl-glycyl-asparagyl-glutaminyl-glutamyl-glutaminyl-valyl-seryl-prolyl-leucyl-threonyl-leucyl-leucyl-lysyl-lysyl-tryptophyl-cysteinyl-Alexa Fluoro 680 C2C2-maleimide conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (panitumumab, 111In-panitumumab, SPECT/CT, surgery) (Experimental): Patients receive loading dose of panitumumab IV over 15 minutes followed by 111In-panitumumab IV bolus on day 0. Patients then undergo SPECT/CT scan between day 1 and day of standard of care surgery (up to day 5). During standard of care surgery, patients receive local injection of optical dye per surgeon's preference and undergo intraoperative and NIR imaging. Patients additionally undergo blood sample collection during screening and ECG during screening, on day 0, and on day 15 if indicated.
  Interventions: Biological: Panitumumab; Other: Indium In 111 Panitumumab; Procedure: Single Photon Emission Computed Tomography; Procedure: Computed Tomography; Procedure: Surgical Procedure; Other: Imaging agent; Procedure: Intraoperative Imaging; Procedure: Near Infrared Imaging; Procedure: Electrocardiography; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Panitumumab — Given by IV
Other: Indium In 111 Panitumumab — Given by IV
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
Procedure: Computed Tomography — Undergo SPECT/CT
Procedure: Surgical Procedure — Undergo standard of care surgery
Other: Imaging agent — Receive local injection of optical dye
Procedure: Intraoperative Imaging — Undergo Intraoperative Imaging
Procedure: Near Infrared Imaging — Undergo Near Infrared Imaging
Procedure: Electrocardiography — Undergo Electrocardiography
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This phase I trial tests the safety and effectiveness of indium In 111 panitumumab (111In-panitumumab) for identifying the first lymph nodes to which cancer has spread from the primary tumor (sentinel lymph nodes) in patients with head and neck squamous cell carcinoma (HNSCC) undergoing surgery. The most important factor for survival for many cancer types is the presence of cancer that has spread to the lymph nodes (metastasis). Lymph node metastases in patients with head and neck cancer reduce the 5-year survival by half. Sometimes, the disease is too small to be found on clinical and imaging exams before surgery. 111In-panitumumab is in a class of medications called radioimmunoconjugates. It is composed of a radioactive substance (indium In 111) linked to a monoclonal antibody (panitumumab). Panitumumab binds to EGFR receptors, a receptor that is over-expressed on the surface of many tumor cells and plays a role in tumor cell growth. Once 111In-panitumumab binds to tumor cells, it is able to be seen using an imaging technique called single photon emission computed tomography/computed tomography (SPECT/CT). SPECT/CT can be used to make detailed pictures of the inside of the body and to visualize areas where the radioactive drug has been taken up by the cells. Using 111In-panitumumab with SPECT/CT imaging may improve identification of sentinel lymph nodes in patients with head and neck squamous cell cancer undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety of indium In 111 panitumumab (111In-panitumumab) as a molecular imaging agent in patients with HNSCC.

SECONDARY OBJECTIVE:

I. Compare sensitivity and specificity of identifying sentinel lymph nodes by systemic injection of 111In-panitumumab prior to day of surgery versus conventional local injection with an optical dye at the time of surgery.

EXPLORATORY OBJECTIVES:

I. Determine if systemic injection of 111In-panitumumab can identify tumor-positive lymph nodes on preoperative SPECT/CT.

II. When preoperative imaging information (eg, fludeoxyglucose F 18 [18F-FDG] positron emission tomography [PET]/CT and/or magnetic resonance imaging [MRI]) data is available:

IIa. Evaluate the sensitivity, specificity, and negative predictive value of 111In-panitumumab SPECT/CT findings to the sensitivity, specificity, and negative predictive value of preoperative MRI in identifying metastatic lymph nodes (histopathological results will serve as the gold standard).

IIb. Evaluate the sensitivity, specificity, and negative predictive value of 111In-panitumumab SPECT/CT findings to the sensitivity, specificity, and negative predictive value of preoperative 18F-FDG PET/CT in identifying metastatic lymph nodes (histopathological results will serve as the gold standard).

OUTLINE:

Patients receive loading dose of panitumumab intravenously (IV) over 15 minutes followed by 111In-panitumumab IV bolus on day 0. Patients then undergo SPECT/CT scan between day 1 and day of standard of care surgery (up to day 5). During standard of care surgery, patients receive local injection of optical dye per surgeon's preference and undergo intraoperative and near infrared (NIR) imaging. Patients additionally undergo blood sample collection during screening and electrocardiography (ECG) during screening, on day 0, and on day 15 if indicated.

Patients are followed for up to 15 days after last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years.
* Biopsy-confirmed diagnosis of squamous cell carcinoma of the head and neck, clinically-staged as node-negative (cN0) or as clinically-suspicious node(s).
* Subjects diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection. Subjects with recurrent disease or a new primary will be allowed.
* Planned standard of care elective neck dissection for node-negative or node-positive disease.
* Have acceptable hematologic status, kidney function, and liver function including the following clinical results:

  * Hemoglobin ≥ 9 gm/dL
  * White blood cell count > 3000/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Serum creatinine ≤ 1.5 times upper reference range

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment.
* History of infusion reactions to monoclonal antibody therapies
* History of allergies to iodine
* Pregnant or breastfeeding.
* Magnesium or potassium lower than the normal institutional values.
* Subjects receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis.
* Severe renal disease or anuria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events grade 2 or higher | Up to 15 days after administration of study drug
  Toxicity graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Summarized by grade, severity and type

SECONDARY OUTCOMES:
Sensitivity of systemic injection of indium In 111 panitumumab (111In-panitumumab) for identifying sentinel lymph nodes | Up to five years
  Will compare the sensitivity of systemic injection of 111In-panitumumab for identifying sentinel lymph nodes to the sensitivity of conventional local injection with an optical dye at the time of surgery. Means and standard deviations for continuous characteristics will be presented. Frequency statistics will be presented for categorical variables. Graphical tools may be used to assess distributional properties of continuous variables.
Specificity of systemic injection of 111In-panitumumab for identifying sentinel lymph nodes | Up to five years
  Will compare the specificity of systemic injection of 111In-panitumumab for identifying sentinel lymph nodes to the sensitivity of conventional local injection with an optical dye at the time of surgery. Means and standard deviations for continuous characteristics will be presented. Frequency statistics will be presented for categorical variables. Graphical tools may be used to assess distributional properties of continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT05901545/ICF_000.pdf